CLINICAL TRIAL: NCT03105765
Title: Effects of Prophylactic Administration of Ketamine on Acute and Chronic Pain After Thoracotomy for Lung Cancer, a Double Blind Randomised Trial.
Brief Title: Acute and Chronic Pain, Especially Neuropathic Pain, After Thoracotomy and Continuous Application of Ketamine.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSK007
Record Dates: First submitted 2016-08-12; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Acute Pain; Chronic Pain; Neuropathic Pain
Keywords: Neuropathic Pain; Chronic Pain; Posterolateral thoracotomy
MeSH Terms: conditions — Acute Pain; Chronic Pain; Neuralgia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): The patients in this Group underwent General anaesthesia with total intravenous anaesthesia containing remifentanil (0,02-0,04 mg/kg ideal Body weight), propofol (4-6 mg/kg ideal Body weight) and atracurium.
  Ketamine 0,2 mg/kg ideal Body weight per hour for 24 hours.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): The patients in this Group underwent General anaesthesia with total intravenous anaesthesia containing remifentanil (0,02-0,04 mg/kg ideal Body weight), propofol (4-6 mg/kg ideal Body weight) and atracurium.
  Placebo (normal Saline) for 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Normal saline applied by bolus before operation started, followed by a continuous application of normal saline for 24 hours.
  Arms: Placebo
Drug: Ketamine — Application of Ketamine 0,2mg/kg ideal Body weight by Bolus before the Operation started, followed by application of 0,2 mg/kg ideal Body weight for 24 hours.
  Arms: Ketamine

SUMMARY:
Chronic Pain, especially neuropathic pain, are adverse events after posterolateral thoracotomy for lung resection. The continuous application of ketamine may have a prophylactic effect and helps to prevent chronic pain. The investigators record the incidence and severity of acute pain and neuropathic pain during a seven day period after thoracotomy as well as the incidence of chronic pain and neuropathic pain after one and three month period. Parallel Group design, comparing one Group with a continuous application (24 hours) of ketamine against a Placebo Group.

ELIGIBILITY:
Inclusion Criteria:

* posterolateral thoracotomy for lung parenchyma resection
* informed consent
* ASA (American Society of Anesthesiologists) Status I-III

Exclusion Criteria:

* history of chronic pain
* history of neuropathic pain
* pregnancy or breastfeeding
* participation in another trial
* hypersensitivity for ketamine
* medication with can influence neuropathic pain (gabapentin, clonazepam)
* history of neurological or behavioral illness
* history of alcohol abuse
* history of chemotherapy or radiation
* opioid medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in perioperative opioid consumption | seven days after operation
  The patients consumption of opioids is recorded once a day for a period of 7 days after operation.
Change in acute pain | 7 days after Operation
  The incidence and severity of pain will be measured using a numeric analog scale (NAS) once a day for a period of seven days after Operation.
acute neuropathic pain | 7 days after operation
  The incidence of neuropathic pain will be measured using the LANSS Pain Scale (Leeds assessment of neuropathic symptoms and signs) three and seven days after operation

SECONDARY OUTCOMES:
Change in chronic Pain | one and three month after operation
  The incidence and severity of pain will be measured using a numeric analog scale (NAS). Pain scale is requested by phone one and three month after Operation.
Chronic Neuropathic pain | one month after operation
  The incidence of neuropathic pain will be measured by using the LANSS Pain Scale (Leeds assessment of neuropathic symptoms and signs) one month after operation
Chronic Neuropathic Pain | three month after operation
  The incidence of neuropathic pain will be measured by using the LANSS Pain Scale (Leeds assessment of neuropathic symptoms and signs) three month after operation
recovery time | eye opening after stopping anesthesia in minutes
  Time between stopping intravenous anaesthesia and first eye opening of the Patient in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Horst Schmidt Klinik, Wiesbaden, Hesse, Germany

REFERENCES:
- [Derived] Ghezel-Ahmadi V, Beck G, Bolukbas S, Ghezel-Ahmadi D. Perioperative ketamine to reduce and prevent acute and chronic post-thoracotomy pain: a randomized, double-blind, placebo-controlled clinical trial. J Thorac Dis. 2024 Dec 31;16(12):8461-8471. doi: 10.21037/jtd-24-648. Epub 2024 Dec 28. PMID 39831260